CLINICAL TRIAL: NCT00990899
Title: Hypertension and Sleep Disordered Breathing in Pediatrics
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 08025
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Hypertension; Obstructive Sleep Apnea
Keywords: hypertension; obstructive sleep apnea; pediatrics
MeSH Terms: conditions — Hypertension; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary objective is to determine the prevalence of sleep disordered breathing in children with primary hypertension or pre hypertension. The secondary objectives are to determine any association factors for children with primary hypertension or prehypertension to have sleep disordered breathing be it gender, age, body mass index (BMI), family history (hx) or ethnic group.

DETAILED DESCRIPTION:
This is an exploratory, cross sectional study involving identification of the children of the age between 10 years and 17 years diagnosed with primary hypertension who have not been previously diagnosed and or treated for sleep disordered breathing with the revised pediatric sleep questionaire (PSQ) for sleep disordered breathing. The subjects that have shown interest will be mailed the informed consent/assent form to tbe reviewed. The consent/assent form will be handed to the child and all their questions and concerns will be answered in a comprehensible manner.

ELIGIBILITY:
Inclusion Criteria:

* aged 10 to 17 years old diagnosed with primary hypertension

Exclusion Criteria:

* refused to participate in the study
* children to secondary hypertension
* previously diagnosed with sleep disordered breathing

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children aged 10 to 17 years who have been diagnosed with primary hypertension
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2008-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melodi Pirzada, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States